CLINICAL TRIAL: NCT00610116
Title: Electronic Repositioning With Acuity and Easytrak Leads
Acronym: ERACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C007-CL-106002
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LV lead electronically repositioning (Other): Single arm study
  Interventions: Device: Electronic Repositioning

INTERVENTIONS:
Device: Electronic Repositioning — Change of pacing vectors for CRT pacing

SUMMARY:
Evaluate appropriate performance of Electronic Repositioning™ (ER) in the clinical routine, cumulative incidence of phrenic nerve stimulation (PNS) & success rates of Electronic Repositioning (ER) to remove it, various incl. left ventricular pacing (LVP) thresholds and PNS

DETAILED DESCRIPTION:
Bipolar leads for left ventricular pacing (LVP) such as the newly available ACUITY™ or the standard EASYTRAK™ II and EASYTRAK™ III leads from GUIDANT in combination with suitable devices for cardiac resynchronization therapy (CRT) allow for the non-invasive programming of different Left Ventricular Pacing (LVP) configurations. Hence, this Electronic Repositioning (ER) may help physicians to overcome problems in cardiac resynchronization therapy (CRT) such as ineffective biventricular pacing, high Left Ventricular Pacing (LVP) thresholds and phrenic nerve stimulation (PNS) without the need for an additional patient's operation to reposition LV leads. The ERACE study it a multi-center, prospective, non-randomized clinical study to document and evaluate appropriate performance of GUIDANT's Electronic Repositioning™ in the clinical routine with respect to the following major aspects:

avoidance of PNS and low LVP thresholds (for low battery consumption and extended device longevity) in standard cardiac resynchronization therapy (CRT)

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving their FIRST implantation of a Left Ventricular (LV) lead in combination with a CRT device with implantable cardioverter defibrillator (ICD) backup and the possibility for Electronic Repositioning™
* Patients willing (= signed written consent) and capable to participate in all procedures of the study"

Exclusion Criteria:

* Patients who will not be available for routine Follow up
* 18 years old
* Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Düsseldorf, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- LV Lead Electronically Repositioning: Single arm study: Electronic Repositioning: Change of pacing vectors for cardiac resynchronization therapy pacing
Period: Overall Study
Arm/Group | LV Lead Electronically Repositioning
Started | 305
Completed | 292 (Number of analyzable patients)
Not Completed | 13

BASELINE CHARACTERISTICS:
Groups:
- LV Lead Electronically Repositioning: Single arm study
  Electronic Repositioning: Change of pacing vectors for Cardiac Resynchronization Therapy pacing
Arm/Group | LV Lead Electronically Repositioning
Number analyzed (Participants) | 292
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 240
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Without the Occurrence of Cardiac Resynchronization Therapy (CRT)-Induced Phrenic Nerve Stimulation (PNS) Between Implant and First Regular Follow-up (FU)
Description: The primary endpoint was the percentage of patients in whom PNS induced by Left Ventricular (LV) pacing could be avoided by electronic repositioning from implantation to first regular follow up (3-6 months postimplant). In this evaluation, prevention of PNS was defined as PNS appearing with the standard pacing configuration-LV tip as cathode versus Right Ventricle (RV) coil as anode-and being avoided by at least one of the three alternative reprogrammable configurations.
Time Frame: From implant until first follow up (occurred between 3 or 6 month after implant procedure)
Measure: Number; unit: participants
Groups:
- Inducible PNS @ Max Output 7V / 0.5 ms: Patients presenting PNS at implant and subsequent follow up (between 3 and 6 months after implant)
Arm/Group | Inducible PNS @ Max Output 7V / 0.5 ms
Number analyzed (Participants) | 292
participants
  Inducible PNS before Electronic Reprogramming | 94
  Remaining PNS after Electronic Reprogramming | 6

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | LV Lead Electronically Repositioning
All-Cause Mortality (participants affected / at risk) | 10/292
Serious Adverse Events (participants affected / at risk) | 40/292
Other Adverse Events (participants affected / at risk) | 32/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LV Lead Electronically Repositioning (N=292)
Pericardial effusion (Cardiac disorders) | 3 (3)
Multiple heart failure symptoms (Cardiac disorders) | 10 (10)
Deep vein thrombosis (DVT) (Cardiac disorders) | 1 (1)
Death (no details) (General disorders) | 5 (5)
Coronary Sinus Dissection (Surgical and medical procedures) | 1 (1)
Gastrointestinal disease (Gastrointestinal disorders) | 1 (1)
Inappropriate pulse generator Shock (Product Issues) | 2 (2)
Increase of Pacing Threshold (Product Issues) | 1 (1)
Ineffective Pulse Generator Shock (Product Issues) | 1 (1)
Inguinal Hernia (Skin and subcutaneous tissue disorders) | 1 (1)
Lead Dislodgment (Product Issues) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pocket hematoma (Product Issues) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Syncope - Non cardiovascular (General disorders) | 1 (1)
Thoracic discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Lead Replacement - Unknown reason (Product Issues) | 1 (1)
Intervention for Coronary Artery Disease (Cardiac disorders) | 2 (2)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1)
Death - Sepsis (Infections and infestations) | 1 (1)
Death - Hemorrhage (Gastrointestinal disorders) | 1 (1)
Death - Heart Failure (Cardiac disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LV Lead Electronically Repositioning (N=292)
Elevated Defibrillation Threshold (Product Issues) | 1 (1)
Elevated Pacing threshold (Product Issues) | 3 (3)
Extracardiac stimulation (Product Issues) | 2 (2)
Pericardial effusion (Cardiac disorders) | 3 (3)
Multiple heart failure symptoms (Cardiac disorders) | 1 (1)
Immunotheraphy (Immune system disorders) | 1 (1)
Atrial Arrhythmia (Cardiac disorders) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (General disorders) | 1 (1)
Cholecystomy (Gastrointestinal disorders) | 1 (1)
Coronary sinus dissection (Surgical and medical procedures) | 1 (1)
Lead Dislodgment (Product Issues) | 5 (5)
Pacing system infection (Product Issues) | 1 (1)
Pocket Hematoma (Product Issues) | 5 (5)
Sepsis (Infections and infestations) | 1 (1)
Pulse Generator system issue (Product Issues) | 1 (1)
Lead - Procedure (Surgical and medical procedures) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No